CLINICAL TRIAL: NCT06613841
Title: Pilot Study to Evaluate Multitracer [18F]Fluciclovine and 18F-FDG PET, and Advanced MRI Methods at 7Tesla Metabolic Profiling of Glioblastoma
Brief Title: Multitracer [18F]Fluciclovine and 18F-FDG PET, and Advanced MRI for Metabolic Profiling of Glioblastoma
Acronym: GBM
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Ali Nabavizadeh, Principal Investigator, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC15324
Record Dates: First submitted 2024-08-28; First posted 2024-09-26 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-05

CONDITIONS: Glioblastoma; Recurrent Glioblastoma; Glioblastoma Multiforme of Brain
Keywords: Early Phase 1; Cohort; Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — fluciclovine F-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Imaging Cohort (Experimental): Up to 15 subjects will enroll in this imaging study at the University of Pennsylvania. Those with a diagnosis of a new intra-axial brain mass that is consistent with GBM per the opinion of a Penn neuroradiologist OR New contrast-enhancing lesion or lesions showing increased enhancement (>25% increase) in a patient with a historical diagnosis of glioblastoma.
  Interventions: Drug: Fluciclovine F18

INTERVENTIONS:
Drug: Fluciclovine F18 — To perform metabolic phenotyping of treatment naïve and recurrent GBM by multitracer [18F]Fluciclovine and 18F-FDG PET.

SUMMARY:
* To perform metabolic phenotyping of treatment naïve and recurrent GBM by multitracer [18F]Fluciclovine and 18F-FDG PET.
* To compare uptake measures of 18F-Fluciclovine and 18F-FDG and MRI quantification of glutamate and lactate levels to tumor tissue laboratory assays (RNA seq and proteomics) of glutamine/glutamate, glucose, and lactate metabolism.
* To perform metabolic phenotyping of treatment naïve and recurrent GBM by advanced MRI methods at 7 Tesla

DETAILED DESCRIPTION:
Subjects with a new intra-axial brain mass that is consistent with glioblastoma (GBM) on brain MRI or post-treatment histologically or molecularly proven GBM who are suspected to have progression and are candidates for surgical resection according to standard of care may be eligible for this study.

Subjects will undergo approximately 45 minutes of dynamic PET/CT scanning after injection of 2 mCi (±20%) of 18F-Fluciclovine. The subject will have a 60-minute break after this initial scan session, they will be allowed to get off the scanner during this time and encouraged to stay hydrated and void as necessary. To confirm that the blood sugar is not high, a glucose test will be performed before the next scan. Subsequently, the subjects will undergo injection of up to 10 mCi of 18F-FDG followed by a static 20-minute scan approximately 60 minutes post injection Subjects will have the option to undergo PET/CT imaging with 18F-Fluciclovine and 18F-FDG on separate days as long as the imaging happens within 7 business days. An optional 60-minute brain MRI without contrast will also be performed with the 7.0 Tesla MRI machine. The timing of the optional second PET scans will be within 7 business days of the baseline PET scans.

Positron emission tomography (PET/CT) imaging will be used to evaluate 18F-fluciclovine and 18F-FDG uptake in treatment naïve and recurrent GBM. Brain MR with Chemical Exchange Saturation Transfer (CEST) and MR spectroscopy (MRS) will be used to determine the glutamate and lactate levels. In addition, clinical brain MRI with and without contrast will be used to evaluate the tumor pre-operatively. This is a non-therapeutic trial in that imaging will not be used to direct treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be ≥ 18 years of age

Must meet the following criteria:

-Diagnosis of a new intra-axial brain mass that is consistent with GBM per the opinion of a Penn neuroradiologist.

OR

* New contrast-enhancing lesion or lesions showing increased enhancement (>25%increase) in a patient with a historical diagnosis of glioblastoma (histologic or molecular proof) on standard MRI after completion of treatment
* Recommended for clinically indicated surgical resection
* Life expectancy of greater than 3 months in the opinion of an investigator or treating physician.
* Karnofsky performance status ≥ 60 per medical record review
* Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

* Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
* Females who are pregnant or breastfeeding at the time of screening will not be eligible for this study; a urine pregnancy test will be performed in women of childbearing potential prior to injection.
* Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study
* Contraindications to MRI
* Only individuals (aged 18 or over) who can understand and give informed consent will be approached to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Uptake Values (SUV) | 2 years
  Quantification of [18F]Fluciclovine and 18F-FDG uptake values (SUV) in treatment naïve and recurrent GBM.

OTHER OUTCOMES:
PET uptake values relation to kinetic parameters | 2 years
  Correlation of PET uptake values (SUV) and kinetic parameters (volume of distribution) with gene expression of glutamine and glucose metabolism.
Quantification of glutamate and lactate levels | 2 years
  The amount of metabolic markers (e.g., glutamate, 5 to 15 mM in normal brain tissue) using 7T MRI. Tumors with high glutamate secretion are associated with increased tumor cell invasiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Nabavizadeh, MD, Principal Investigator — University of Pensylvania
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Nabavizadeh A, Bagley SJ, Doot RK, Ware JB, Young AJ, Ghodasara S, Zhao C, Anderson H, Schubert E, Carpenter EL, Till J, Henderson F Jr, Pantel AR, Chen HI, Lee JYK, Amankulor NM, O'Rourke DM, Desai A, Nasrallah MP, Brem S. Distinguishing Progression from Pseudoprogression in Glioblastoma Using 18F-Fluciclovine PET. J Nucl Med. 2023 Jun;64(6):852-858. doi: 10.2967/jnumed.122.264812. Epub 2022 Dec 22. PMID 36549916